CLINICAL TRIAL: NCT00017966
Title: Cortical Excitability During Self-Paced Voluntary Movements
Brief Title: Brain Excitability During Self-Paced Voluntary Movements
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010199; 01-N-0199
Record Dates: First submitted 2001-06-23; First posted 2001-06-25 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Movement Disorder; Healthy
Keywords: Transcranial Magnetic Stimulation; Motor Cortex; Cerebral Inhibition; Corpus Callosum; Evoked Potential; Healthy Volunteer; Normal Control
MeSH Terms: conditions — Movement Disorders

SUMMARY:
This study will use transcranial magnetic stimulation to examine how the brain controls movement by sending messages to the spinal cord and muscles and what goes wrong with this process in disease. Normal healthy volunteers 18 years of age and older may be eligible to participate.

In transcranial magnetic stimulation, an insulated wire coil is placed on the subject's scalp or skin. Brief electrical currents are passed through the coil, creating magnetic pulses that stimulate the brain. During the stimulation, participants will be asked to tense certain muscles slightly or perform other simple actions. The electrical activity of the muscle will be recorded on a computer through electrodes applied to the skin over the muscle. In most cases, the study will last less than 3 hours.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the influence of volitional movement on excitability of ipsilateral as well as contralateral motor cortical neurons controlling homologous and surrounding muscles. Transcallosal and surrounding inhibitions are well known phenomenon to suppress unwanted movements during voluntary action, which is often disturbed in various movement disorders. Transcranial magnetic stimulation (TMS) has been used to investigate these inhibitory mechanisms, but the inhibitory influence during and after voluntary movement has not been well elucidated yet. In normal volunteers, we plan to determine if voluntary movements of one finger influence the cortical excitability responsible for surrounding as well as contralateral homologous muscles, using voluntary movement-triggered TMS. The primary outcome measures would be any changes in motor evoked potential (MEP) size and intracortical inhibition (ICI) parameters.

ELIGIBILITY:
Normal adult volunteers 18 or more years old.

Subjects must not have medico-surgical illness.

Subjects must not have neurological illness.

Subjects must not have psychiatric illness.

Subjects must not be taking any medication with potential influence on nervous system function.

Subjects must not have a pacemaker.

Subject must not have an implanted medical pump.

Subjects must not have a metal plate or a metal object in the skull or eye.

Subjects must not have a history of seizure disorder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2001-06; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Blakemore C, Carpenter RH, Georgeson MA. Lateral inhibition between orientation detectors in the human visual system. Nature. 1970 Oct 3;228(5266):37-9. doi: 10.1038/228037a0. No abstract available. PMID 5456209
- [Background] Prince DA, Wilder BJ. Control mechanisms in cortical epileptogenic foci. "Surround" inhibition. Arch Neurol. 1967 Feb;16(2):194-202. doi: 10.1001/archneur.1967.00470200082007. No abstract available. PMID 6018049
- [Background] Krnjevic K. Role of GABA in cerebral cortex. Can J Physiol Pharmacol. 1997 May;75(5):439-51. No abstract available. PMID 9250378